CLINICAL TRIAL: NCT03787823
Title: Robotic Retzius-sparing Radical Prostatectomy- a Randomized Controlled Trial Evaluating Transdouglas-RARP
Brief Title: RCT-evaluation of Retzius-sparing Robotic Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Joanne N. Nyarangi-Dix, M.D., Chief senior physician and Vice chairlady of the Dept. of Urology, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Transdouglas RCT-Study
Record Dates: First submitted 2018-09-04; First posted 2018-12-26 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retzius-sparing RARP (Other): Arm B randomizes men with an indication for radical robotic Prostatectomy (RARP) to retzius-sparing transdouglas RARP
  Interventions: Procedure: robotic Prostatectomy (RARP)
- anterior transperitoneal RARP (Other): Arm A randomizes men with an indication for radical robotic Prostatectomy (RARP) to anterior transperitoneal RARP
  Interventions: Procedure: robotic Prostatectomy (RARP)

INTERVENTIONS:
Procedure: robotic Prostatectomy (RARP) — Modification of robotic Prostatectomy Arm A classic technique/ anterior transperitoneal RARP Arm B Transdouglas Technique/retzius-sparing RARP

SUMMARY:
Prospective randomized blinded RCT comparing Transdouglas Prostatectomy to classical transperitoneal anterior radical prostatectomy

DETAILED DESCRIPTION:
We will evaluate functional urinary and sexual recovery, oncologic outcomes and postoperative complications in patients over a follow up period of 12 months

ELIGIBILITY:
Inclusion Criteria:

* Indication for radical prostatectomy
* >18 years old
* Literate
* Preoperatively continent
* informed signed consent for study

Exclusion Criteria:

* cT4-Cancer
* Withdrawl of consent to study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 186 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Urinary continence | 1 Week after Prostatectomy
  Pad use

SECONDARY OUTCOMES:
Resection margine | pathology report, approximately 1 week postoperatively
Urinary continence | 3, 6 and 12 months after Prostatectomy
  Pad use
Postoperative complications | First 12 months after Prostatectomy
postoperative PSA | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
So far, no sharing planed